CLINICAL TRIAL: NCT05775055
Title: A Comparison of Three Commercial Oral Rehydration Solutions Consumed After Extra-cellular Dehydration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: entrinsic bioscience LLC (Unknown)
Responsible Party: Principal Investigator, Lewis James, Reader in Nutrition, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LEON8472
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Fluid Balance Outcomes

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, crossover design
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Commercially Available Oral Rehydration Solution A (Experimental): A commercially available oral rehydration solution (~2.8% carbohydrate, ~45 mmol/L sodium, ~20 mmol/L potassium, 34 mmol/L chloride)
  Interventions: Other: Composition of oral rehydration solutions
- Commercially Available Oral Rehydration Solution B (Experimental): A commercially available oral rehydration solution (~0.1% carbohydrate, ~2% amino acids (protein), ~67 mmol/L sodium, ~20 mmol/L potassium, 30 mmol/L chloride)
  Interventions: Other: Composition of oral rehydration solutions
- Commercially Available Oral Rehydration Solution C (Experimental): A commercially available oral rehydration solution (~2.2% carbohydrate, ~45 mmol/L sodium, ~20 mmol/L potassium)
  Interventions: Other: Composition of oral rehydration solutions

INTERVENTIONS:
Other: Composition of oral rehydration solutions — Investigate the efficacy of an amino acid-based oral rehydration solution compared to two current commercially available glucose-based oral rehydration solutions.

SUMMARY:
Dehydration is commonplace in a number of settings, including exercise, daily living (i.e. inadequate fluid intake) and with relatively common bacterial/viral infections that induce diarrhoea and/or vomiting. As such, it is important to develop effective strategies to facilitate the recovery and maintenance of body water (i.e. rehydration). Whilst rehydration from exercise dehydration has been well-studied, rehydration from other types of dehydration have not. Despite this, oral rehydration solutions have been produced and are commercially available (in chemists/pharmacies and supermarkets) to help recover from dehydration produced by illnesses like diarrhoea and vomiting. Most commercially available oral rehydration solutions use a sugar-base (glucose) and a mixture of electrolytes, but little work has gone into evaluating the efficacy of such solutions. Furthermore, more recent work has explored the use of proteins that they may offer some advantage over sugar/glucose-based beverages.

Therefore, the aim of this study is to investigate the efficacy of a protein-based oral rehydration solution compared to two current commercially available glucose-based oral rehydration solutions.

DETAILED DESCRIPTION:
Dehydration refers to a decrease in body water and occurs when water losses in urine, sweat or other body fluid secretions (e.g vomit or diarrhoea) exceed fluid intake in drinks and foods. Indeed, dehydration is commonplace in a number of settings, including exercise, daily living (i.e. inadequate fluid intake) and with relatively common bacterial/viral infections that induce diarrhoea and/or vomiting. As such it is important to develop effective strategies to facilitate the recovery and maintenance of body water (i.e. rehydration).

Whilst rehydration from exercise dehydration has been well-studied, rehydration from other types of dehydration have not. Despite this, oral rehydration solutions have been produced and are commercially available (in chemists/pharmacies and supermarkets) to help recover from dehydration produced by illnesses like diarrhoea and vomiting. Oral rehydration solutions have been developed that vary in their composition for both electrolytes and other nutrients (glucose, amino acids etc.). Most commercially available oral rehydration solutions use a sugar-base (glucose) and a mixture of electrolytes, but little work has gone into evaluating the efficacy of such solutions. Furthermore, more recent work has explored the use of amino acids (the building blocks of proteins) in isolation or as complete proteins and suggest that they may offer some advantage over sugar/glucose-based beverages.

Dehydration produced by illnesses like diarrhoea and vomiting cause water an electrolyte losses that are different in nature to exercise and as such, exercise is not a good way to study these effects. The type of dehydration produced with diarrhoea and vomiting can be mimicked by using a diuretic like furosemide. This type of diuretic is used clinically in situations of water overload (e.g. congestive heart failure or high blood pressure) and are used daily for months in many patients. They produce mild dehydration (~2-2.5%) and thus offer the opportunity to understand recovery from the type of dehydration caused by illness, without the presence of illness.

Given the body water contains high amounts of salts (electrolyte), when dehydration occurs electrolytes are also lost from the body. These electrolytes are needed to retain water in the various spaces of the body (inside cells, in the blood etc.) and thus failure to replace the electrolytes lost during dehydration will lead to a less effective rehydration response. Therefore, commercial oral rehydration solutions contain a balance of different electrolytes to replace those lost with dehydration and to help retain the ingested fluid. However, different formulations use a different balance of electrolytes and little work has examined the efficacy of these different formulations.

Therefore there is a need to understand the efficacy of different oral rehydration solution formulations following dehydration, something that has received little attention to date, surprisingly. Therefore, this study will compare the rehydration efficacy of a commercial amino-acid based oral rehydration solution compared to two current commercially available glucose-based oral rehydration solutions after dehydration induced by a diuretic.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* male or female
* good health

Exclusion Criteria:

* Gastrointestinal, cardiovascular or renal conditions; other health conditions that might influence the study outcomes.
* Medication use (e.g. anti-biotics, diuretics, NSAIDS etc.) that might influence the study outcomes or interact with furosemide.
* Allergy to sulfonamides (sulfa drugs).
* Smoking (including vaping)
* Amenorrhoeic females
* Any high-level/elite athlete, or aspiring high level athlete, where drug testing/regulations are carried out and regulations need to be followed (furosemide is prohibited in sport as it is used as a masking agent).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Net fluid balance | 9 hours
  Determined from urine output and drink volume collected before and after drink ingestion
Drink retention | 4 hours
  Determined from urine output and drink volume collected before and after drink ingestion
Electrolyte balance | 9 hours
  Determined from electrolyte concentrations (i.e., sodium, potassium, chloride) in urine and drink samples before and after drink ingestion
Speed of rehydration | 4 hours
  Determined from urine output and drink volume collected before and after drink ingestion

SECONDARY OUTCOMES:
Plasma volume | 9 hours
  Determined from haemoglobin and haematocrit measures in blood samples collected before and after drink ingestion
Plasma osmolality | 9 hours
  Determined from venous blood samples collected before and after drink ingestion
Urine volume | 9 hours
  Determined from urine samples collected before and after drink ingestion
Urine electrolyte concentration (i.e., sodium, potassium, chloride) | 9 hours
  Determined from urine samples collected before and after drink ingestion
Blood electrolyte concentration (i.e., sodium, potassium, chloride) | 9 hours
  Determined from blood samples collected before and after drink ingestion
Body mass change | 9 hours
  Determined from weighing participants before and after drink ingestion
Urine specific gravity | 9 hours
  Determined from urine samples collected before and after drink ingestion

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No